CLINICAL TRIAL: NCT00305552
Title: Randomized Controlled Trial of Thalidomide vs Placebo in Skin Sarcoidosis
Brief Title: SARCOTHAL. Thalidomide in Skin Sarcoidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Myriem CARRIER, Department Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P031008
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2007-01

CONDITIONS: Sarcoidosis
Keywords: Randomized controlled trial; Thalidomide vs placebo; skin sarcoidosis; Thalidomide
MeSH Terms: conditions — Sarcoidosis | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): THALIDOMIDE
  Interventions: Drug: THALIDOMIDE

INTERVENTIONS:
Drug: THALIDOMIDE — THALIDOMIDE

SUMMARY:
Sarcoidosis is a multisystem disease involving most frequently the lung, the eyes, the lymph nodes and the skin. Skin lesions may be disfiguring and impair the quality of life. Thalidomide is a multi-target drug that has been shown to be of benefit in skin sarcoidosis in case reports. The objective is to assess the efficacy and tolerance of thalidomide in skin sarcoidosis.

DETAILED DESCRIPTION:
The study consists in comparing thalidomide to placebo in skin sarcoidosis. Patients with sarcoidosis not necessitating a high-dose corticosteroid regimen, and assessable skin lesions, are eligible. They are randomized and receive either thalidomide or placebo for 3 months. Then they are given Thalidomide for a 3-month open-label period.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven skin sarcoidosis
* Assessable target skin lesions

Exclusion Criteria:

* Rapidly evolving sarcoidosis
* Patients necessitating a corticosteroid regimen of more than 15mg per day.
* Women not willing to undertake a contraceptive method.
* Neurologic impairment
* Past treatment with Thalidomide
* Renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Size of target skin lesions at 3 months. | during de study
  Size of target skin lesions at 3 months.

SECONDARY OUTCOMES:
Physician global assessment at 3 months. Functional assessment of other organs. Side-effects at 3 months. | during the study
  Physician global assessment at 3 months. Functional assessment of other organs. Side-effects at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michel RYBOJAD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- HOPITAL Saint Louis, Service de Dermatologie, Paris, France

REFERENCES:
- [Derived] Droitcourt C, Rybojad M, Porcher R, Juillard C, Cosnes A, Joly P, Lacour JP, D'Incan M, Dupin N, Sassolas B, Misery L, Chevrant-Breton J, Lebrun-Vignes B, Desseaux K, Valeyre D, Revuz J, Tazi A, Chosidow O, Dupuy A. A randomized, investigator-masked, double-blind, placebo-controlled trial on thalidomide in severe cutaneous sarcoidosis. Chest. 2014 Oct;146(4):1046-1054. doi: 10.1378/chest.14-0015. PMID 24945194